CLINICAL TRIAL: NCT01186172
Title: Lock Con Etanolo Per il Salvataggio di Dispositivi Vascolari a Lungo Termine. Un Trial Clinico Multicentrico Controllato Randomizzato
Brief Title: Ethanol Lock for the Salvage of Infected Long-term Vascular Access
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Michele Pagani, Dirigente Medico 1 livello, Fondazione IRCCS Policlinico San Matteo di Pavia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ETHCVC
Record Dates: First submitted 2010-08-17; First posted 2010-08-23 (Estimated); Last update posted 2012-01-05 (Estimated); Status verified 2012-01

CONDITIONS: Bacteremia
Keywords: ethanol; lock therapy; vascular access; central venous catheter; sepsis
MeSH Terms: conditions — Bacteremia; Sepsis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ethanol-lock (Experimental): Treatment with a combination of ethanol-lock and parenteral therapy
  Interventions: Drug: Ethanol-lock therapy
- Antibiotic lock (Active Comparator): Treatment with a combination of antibiotic-lock and parenteral therapy
  Interventions: Drug: Antibiotic-lock

INTERVENTIONS:
Drug: Ethanol-lock therapy — Daily ethanol-lock with 70% ethanol instilled in device dead-space, leaved in place for the longest possible interval, and then discarded. For dialysis devices, it is acceptable to leave the lock in place between dialysis sessions. Lock therapy will be continued for 7 days.
  Arms: Ethanol-lock
Drug: Antibiotic-lock — Daily antibiotic-lock according to 2009 IDSA Guidelines,instilled in device dead-space, leaved in place for the longest possible interval, and then discarded. For dialysis devices, it is acceptable to leave the lock in place between dialysis sessions. Lock therapy will be continued for 7 days.
  Arms: Antibiotic lock

SUMMARY:
Long-term venous devices (e.g.Ports, tunneled catheters,...) may become infected. Sometimes it is very difficult to treat the infection and it is necessary to remove the device. The purpose of this study is to determine the efficacy of instilled ethanol ("ethanol lock therapy") versus instilled antibiotics ("antibiotic lock therapy") to save long-term venous device when infected, preventing their removal.

ELIGIBILITY:
Inclusion Criteria:

* Age: >1 year and 10 Kgs
* Long-term vascular device in place at least for 7 days
* Catheter-related infection (at least presumed)
* Will to save the infected device (expected high risk access)

Exclusion Criteria:

* Known ethanol-allergy
* Known antabuse-like drugs in use
* Religious refusal
* S.aureus or Candida spp. as main pathogens (except in the unusual and documented scenarios when replacement of vascular access device proved to be very difficult)
* Tract or pocket infection
* Complicated infection (septic shock, infectious thrombosis, osteomyelitis, endocarditis)

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2010-06; Primary Completion 2012-12 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Ratio of saved devices | 7 days

SECONDARY OUTCOMES:
Number of participants with adverse events linked to ethanol lock as a measure of safety and tolerability | 60 days
  Major adverse event (stop protocol): anaphylaxis, antabuse-like reaction, device damage, severe dysphoric reaction.
  Minor adverse events (do not stop protocol): nausea, vomiting, headache, dizziness.
Number of patients with proper parenteral therapy | 7 days
  Verified by an Infectious Diseases Specialist
Ratio of saved devices | 15-30-60 days
Time for next bacteriemic episode | 30 days after the end of lock

CONTACTS AND LOCATIONS:
Overall Officials: Michele Pagani, M.D., Principal Investigator — Fondazione IRCCS Policlinico San Matteo, Pavia, Italy
Locations (1):
- Fondazione IRCCS Policlinico "San Matteo", Pavia, PV, Italy

REFERENCES:
- [Background] Maiefski M, Rupp ME, Hermsen ED. Ethanol lock technique: review of the literature. Infect Control Hosp Epidemiol. 2009 Nov;30(11):1096-108. doi: 10.1086/606162. PMID 19803767